CLINICAL TRIAL: NCT00696319
Title: Dynamic Stability of the ACL Deficient Knee - a Prospective Cohort Study
Brief Title: Dynamic Stability of the Anterior Cruciate Ligament (ACL) Deficient Knee
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was suspended due to lack of resources.
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Delaware (Other)
Responsible Party: May Arna Risberg, PT, PhD, NAR/Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-2008-NAR; NIH grant #2RO1HD37985-05
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Knee Injury
Keywords: Rupture of the anterior cruciate ligament of the knee
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Arm 1 will go through a rehabilitation protocol with perturbation training exercises.
  Interventions: Other: Exercise protocol with perturbation exercises.
- 2 (Experimental): Arm 2 will go through a rehabilitation protocol with traditional exercises for balance and stability training.
  Interventions: Other: Exercise protocol with traditional exercises for stability and balance.

INTERVENTIONS:
Other: Exercise protocol with perturbation exercises. — Perturbation exercises are exercises for balance and stability that involves perturbations of the surface through use of custom made equipment (a rollerboard, a rockerboard and a platform).
  Arms: 1
Other: Exercise protocol with traditional exercises for stability and balance. — The exercise protocol will consist of exercises for balance and stability that do not include sudden disturbances or perturbations to the surface.
  Arms: 2

SUMMARY:
The study that is registered in ClinicalTrials is a part study of an overall study with the title 'Dynamic stability of the ACL-injured knee'. The aim of the overall study is to prospectively follow a cohort of newly injured patients with total rupture of the anterior cruciate ligament in the knee, in order to document results from different rehabilitation regimes after the injury.

The title of the part study is 'Neuromuscular changes in ACL-deficient individuals before and after an intensive perturbation training program. A case-control study.' The aims of the part study are:

1. To describe muscle activation patterns, joint angles and forces during gait and one-legged hop in newly injured ACL-deficient individuals before and after execution of an intensive training program consisting of either perturbation training or conventional balance- and stability training
2. To describe eventual changes between the two groups that may indicate superiority of either one of the methods

The study will include 25 subjects in each group. The intervention consists of two different rehabilitation protocols for neuromuscular training. Subjects will be tested in a biomechanical laboratory before and after intervention, with use of 3D camera systems, force plates and electromyographic measurements (EMG). Main outcomes are eventual differences in muscle activation patterns, joint angles and forces during selected phases of walking and one-legged hopping. Secondary outcomes of interest are self-assessment of knee function, isokinetic strength and functional one-legged hop tests.

Status: Inclusion to the main study started in January 2007. Data collection for the case-control part study will take place in 2008-2009. The part study study should be finished in 2010, where results will be included in a PhD dissertation. The PhD student responsible, Ingrid Eitzen, is enrolled in the Doctoral program at the Faculty of Medicine, University of Oslo. She is employed at Orthopaedic Centre, Ullevaal University Hospital and part of The Norwegian Research Center for Active Rehabilitation (NAR). The project is included in the NAR research program. In addition, the overall study is organized as a formalized collaboration with the University of Delaware, US, where they also will follow a cohort of 150 subjects.

DETAILED DESCRIPTION:
The study 'Dynamic stability of the ACL-injured knee' is carried out as part of a formalized research collaboration between the University of Delaware, US, and NAR, Orthopaedic Centre, Ullevaal University Hospital, Norway. The project is funded by National Institutes of Health. 150 patients, both men and women, aged between 13-55 years, will over a three year-period be enrolled in the study. Follow-up time is 2 years. A part-study will have a case-control design and include 50 of the patients.

In Norway, approximately 4000 persons rupture their anterior cruciate ligament (ACL)per year. The majority of these individuals are relatively young people, engaged in various physical activities. Most ACL-ruptures occur within pivoting sports like soccer, team handball, floorball, basketball and volleyball, but also within racket sports, ice-hockey, dance/gymnastics and alpine skiing. A ruptured ACL is a serious injury for the individual, who often experiences exclusion form both work, leisure activities and sports for potentially a long period of time. A considerable number of the patients will not be able to return to their pre-injury activity level, and many will also experience long time consequences, the most serious of these being development of knee osteoarthritis(OA).

The function of the injured knee varies considerably among patients with a torn ACL. Some are able to stabilize their knees even during demanding activities and sports, while others experience frequent episodes of giving way, also following daily activities. Currently, there is little consensus regarding the optimal rehabilitation program following ACL injury and/or criteria for ACL-reconstruction. But, whether managed operatively or non-operatively, a full return to pre-injury activities after ACL rupture is always dependent on the development of dynamic knee stability. In the past 10-15 years, a test battery consisting of standardised and validated tests for screening and classification of newly injured ACL-patients has been developed. The test battery includes four different functional one-legged hop tests, two questionnaires on knee function and self-evaluation of knee status in the form of a global rating. The questionnaires included are The Knee Outcome Survey - Activities of Daily Living (KOS-ADL), and The International Knee Documentation Subjective Knee Form (IKDC 2000). In addition, we measure the laxity between the tibia and femur with KT1000, register eventual number of episodes of giving way and perform isokinetic strength measurements of the quadriceps and hamstrings muscles with a Biodex6000 system. Based on these tests, all newly diagnosed patients with an ACL-rupture may be classified according to whether they have good or poor dynamic stability. Those with 80% or more performance on the injured leg compared to the non-injured leg on all hop tests, who score 80 or more in KOS-ADL, who rate themselves to a score of at least 60 on the global rating and have experienced maximum one episode of giving way, are categorized as potential copers. Those who score below these limits and/or have experienced two or more episodes of giving way are categorized as non-copers. In Norway, approximately 50% of all ACL-injured individuals go through reconstructive surgery. The optimal time to decide whether surgery is the best treatment option or not is highly individual, but recent research has demonstrated that the functional status of the knee at the time of eventual surgery is more important than the time span since the date of injury. Reconstructive surgery will to a large degree re-establish the mechanical stability of the knee, but has not been proven to provide sufficient dynamical stability or make the patient able to return to his/hers pre-injury activity level. It can at present time neither be documented that reconstructive ACL-surgery reduces the risk of later development of knee OA.

Several questions remain that will affect the development of effective rehabilitation programs for patients after ACL rupture. Validated practice guidelines for patients after ACL injury that discriminate between surgical and non-surgical candidates, lead to a return to pre-injury activities, and protect future joint health have not been reported. The case-control part study will aim specifically to investigate the effectiveness of two different protocols for neuromuscular training, with before- and after intervention data collection in a biomechanical laboratory.

Results from the overall study (inclusive the part study) will allow us to extend our previous findings and will provide information that is needed to identify and treat individuals with ACL rupture across the spectrum of compensation strategies.

Follow-up during the project includes

* Functional one-legged hop tests
* Instrumental measurement of knee laxity (KT1000)
* Isokinetic strength testing of the quadriceps and hamstrings muscles
* Biomechanical analyses of gait and one-legged hops in the Motion Analysis Laboratory at the Norwegian University of Sport Sciences
* Self-assessment of knee function in the form of global rating

ELIGIBILITY:
Inclusion Criteria:

* Verified unilateral total rupture of the ACL
* Age 13-55 years
* Date of injury within 3 months prior to inclusion
* Activity level 1 or 2 (regular participation in pivoting sports)

Exclusion Criteria:

* Concomitant ligamentous injury
* Bilateral involvement
* Symptomatic meniscal damage
* Fractures
* Full-thickness articular cartilage damage larger than 1 cm in diameter

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Biomechanical changes during walking and one-legged hop tests. | Before and after a six week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: May Arna Risberg, PT, PhD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Orthopaedic Centre, Ullevaal University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- See also: Related Info — http://active-rehab.no/